CLINICAL TRIAL: NCT06742879
Title: A Multi-center Clinical Study of Zanubrutinib in Combination With First-line Chemoimmunotherapy in Patients With Grade 3A High-risk Follicular Lymphoma
Acronym: ZCM3AHRFL
Status: Active, not recruiting | Type: Observational
Sponsor: Zhengzhou University (Other)
Responsible Party: Principal Investigator, Mingzhi Zhang, Professor, Zhengzhou University
Other Study IDs: 3AHRFL20240901; ZhengZhouU (Other: the first affiliated hospital of zhengzhou university)
Record Dates: First submitted 2024-12-02; First posted 2024-12-19 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2024-12

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Wax blocks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Background： At present, there is controversy about whether FL3a is treated as FL or DLBCL. Relevant studies have shown that compared with patients with FL3a grade 1~2, they have unique immunohistochemical characteristics, and there are some differences in clinical features and outcomes. In patients with FL3a, the Ki-67 index is higher, the recurrence rate is higher, there is more histologic transformation, the prognosis is worse, and the likelihood of lymphoma-related death is higher. Bruton's tyrosine kinase (BTK) is a key kinase in the B-cell signaling pathway, and studies have shown that BTK inhibitors including zanubrutinib combined with traditional immunochemotherapy regimens may have a synergistic effect in the treatment of B-cell malignancies, and the combination has become one of the current clinical research directions.

Aim:

To assess the efficacy and safety of zanubrutinib in combination with first-line immunochemotherapy in high-risk patients with FL3a.

DETAILED DESCRIPTION:
Bruton's tyrosine kinase (BTK) is a key kinase in the B-cell signaling pathway, and its abnormal activation leads to abnormal activation of the B-cell receptor signaling pathway, B-cell malignant proliferation, and lymphoma.

There is controversy about whether FL3a is treated as FL or DLBCL. Relevant studies have shown that compared with patients with FL3a grade 1~2, they have unique immunohistochemical characteristics, and there are some differences in clinical features and outcomes. In patients with FL3a, the Ki-67 index is higher, the recurrence rate is higher, there is more histologic transformation, the prognosis is worse, and the likelihood of lymphoma-related death is higher. Bruton's tyrosine kinase (BTK) is a key kinase in the B-cell signaling pathway, and studies have shown that BTK inhibitors including zanubrutinib combined with traditional immunochemotherapy regimens may have a synergistic effect in the treatment of B-cell malignancies, and the combination has become one of the current clinical research directions.

The recent study is to assess the efficacy and safety of zanubrutinib in combination with first-line immunochemotherapy in high-risk patients with FL3a.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-70 years old (including 18 years old and 70 years old), ECOG score 0-2 points; 2. Confirmed diagnosis of follicular lymphoma with pathological grade of 3A (pathological report of three months before enrollment is acceptable) (Note: If there is any doubt about the pathological diagnosis, a domestic third-party consultation can be organized); 3. Treatment-naïve patients with indications for treatment; 4. Meet at least one of the criteria for high tumor burden in GELF; 5. Have not received other tumor-related treatments in the past; 6. Acceptable hematological indexes, no contraindications to chemotherapy; 7. Liver function: TBIL≤1.5×ULN; ALT or AST ≤2.5×ULN; Alkaline phosphatase ≤3×ULN in patients with non-bone invasion; 8. Renal function: serum creatinine ≤1.5×ULN; 9. Female and male patients of childbearing potential and their spouses are willing to use adequate contraception throughout the study period, and female patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose; 10. Subjects voluntarily participated in the clinical trial, signed the informed consent form, and cooperated with the follow-up.

Exclusion Criteria:

* 1. Refusal to collect blood specimens; 2. Previous allergy to any of the medications in the regimen; 3. Pregnant and lactating women; 4. Significant illness that, in the opinion of the investigator, can cause trial interference; 5. Combined with other tumors; 6. Presence of contraindications related to the treatment of the drug in the protocol; 7. Those with severe mental illness; 8. Participating in other clinical trials; 9. Prior treatment with anti-tumor therapy (such as radiotherapy, chemotherapy, hormonal therapy, biological therapy, immunotherapy); 10. Other serious diseases that may limit the subject's participation in this trial, such as: uncontrolled diabetes mellitus; Severe cardiac insufficiency (NYHA classification II or above); Acute coronary syndrome within the past 6 months; Coronary revascularization such as stenting, coronary artery bypass surgery, and other heart and large vessel related surgeries in the past 6 months; Severe arrhythmias include frequent premature ventricular episodes, ventricular tachycardia, rapid atrial fibrillation/atrial flutter, and severe bradycardia. Uncontrolled hypertension: systolic blood pressure > 150 mmHg, diastolic blood pressure > 100 mmHg. Gastric ulcer (gastric ulcer judged by the investigator to be at risk of perforation); Active autoimmune disease (e.g., systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjögren's syndrome, autoimmune thrombocytopenia, etc.); Severe respiratory diseases (such as obstructive pulmonary disease and history of bronchospasm), etc.; 11. In the opinion of the investigators, it is not suitable for enrollment; 12. Hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer test is not within the normal reference value; Those who are positive for hepatitis C virus (HCV) antibody and positive for hepatitis C virus (HCV) RNA in peripheral blood; Those who are positive for human immunodeficiency virus (HIV) antibodies; Those who test positive for syphilis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Age 18-70 years old (including 18 years old and 70 years old), ECOG score 0-2 points; Confirmed diagnosis of follicular lymphoma with pathological grade of 3A; Treatment-naïve patients with indications for treatment; Meet at least one of the criteria for high tumor burden in GELF;Have not received other tumor-related treatments in the past;Acceptable hematological indexes, no contraindications to chemotherapy; Liver function: TBIL≤1.5×ULN; ALT or AST ≤2.5×ULN; Alkaline phosphatase ≤3×ULN in patients with non-bone invasion;Renal function: serum creatinine ≤1.5×ULN;Female and male patients of childbearing potential and their spouses are willing to use adequate contraception throughout the study period, and female patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose;Subjects voluntarily participated in the clinical trial, signed the informed consent form, and cooperated with the follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
CR | 2 years
  complete response

SECONDARY OUTCOMES:
ORR | 2 years
  ORR: the proportion of patients whose tumors shrink by 30% and remain in effect for more than 4 weeks.
PFS of 2 years | 2 years
  PFS of 2 years: the time from the start of treatment to the time when the patient has progressed on the disease or dies due to any cause in 2 years.
OS of 2 years | 2 years
  OS of 2 years: the time from the time when the patient receives treatment to the time when the patient dies due to any cause in 2 years.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of zhengzhou University, Zhengzhou, Henan, China